CLINICAL TRIAL: NCT04837482
Title: Evaluating the Impact of AGN-190584 on Night-driving Performance
Brief Title: A Study to Assess the Impact and Adverse Events of Topical Eyedrops of AGN-190584 on Night-driving Performance in Participants, 40 to 55 Years of Age
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1883-306-013
Record Dates: First submitted 2021-04-06; First posted 2021-04-08 (Actual); Results first posted 2024-10-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-09

CONDITIONS: Presbyopia
Keywords: Presbyopia; AGN-190584
MeSH Terms: conditions — Presbyopia | interventions — Pilocarpine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- AGN-190584 Sequence 1 (Experimental): AGN-190584 Sequence 1 (Participants will receive AGN-190584 from Visit 2 through Visit 3 followed by Vehicle from Visit 4 through Visit 5).
  Interventions: Drug: AGN-190584; Drug: Vehicle
- AGN-190584 Sequence 2 (Experimental): AGN-190584 Sequence 2 (Participants will receive Vehicle from Visit 2 through Visit 3 followed by AGN-190584 from Visit 4 through Visit 5).
  Interventions: Drug: AGN-190584; Drug: Vehicle

INTERVENTIONS:
Drug: AGN-190584 — Topical eyedrop
  Other Names: Pilocarpine hydrochloride, 1.25%
Drug: Vehicle — Topical eyedrop
  Other Names: Pilocarpine HCl Placebo

SUMMARY:
The purpose of this study is to evaluate night-driving performance in real-world driving conditions in participants with presbyopia treated with AGN-190584 versus vehicle. Adverse events and change in disease symptoms will be assessed.

AGN-190584 is an investigational formulation of pilocarpine for treating symptoms associated with presbyopia as a topical, once-daily eyedrop delivered by a proprietary vehicle.

This crossover study consists of two parts. Part 1 consists of Visit 2 and Visit 3, and Part 2 consists of Visit 4 and Visit 5. Approximately half of the participants will receive AGN-190584 at Visit 2 through Visit 3 (Sequence 1 participants) and the remaining participants (Sequence 2 participants) will receive AGN-190584 at Visit 4 through Visit 5. All participants will receive AGN-190584 at home as instructed. Approximately 54 adult participants with presbyopia will be enrolled at 1 site in Australia.

Treatment duration is expected to be no more than 71 days. In Part 1, at Visit 2 (Day 1) and at home as instructed for 7 to 14 days, Sequence 1 participants will receive 1 eyedrop of AGN-190584 in each eye and Sequence 2 participants will receive 1 eyedrop of vehicle in each eye. All participants will have a driving assessment at Visit 3 (Day 8 to 15). In Part 2, at Visit 4 (Day 15 to 57) and at home as instructed for 7 to 14 days, Sequence 2 participants will receive 1 eyedrop of AGN-190584 in each eye and Sequence 1 participants will receive 1 eyedrop of vehicle in each eye. All participants will have a driving assessment at Visit 5 (Day 22 to 71).

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the course of the study at a hospital or clinic. The effects of the treatment will be checked by medical assessments, asking about side effects, and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* In good general health at the screening visit, as determined by the investigator from medical history.
* Subjective complaints of poor near vision that impacts activities of daily living, as defined by at least a moderate impact (score > = 3) on at least 1 question on NEI VFQ-25 Questions 5 to 7 in the main questionnaire or near vision subscale, Questions A3 to A5 in the Appendix of Optional Additional Questions, at the screening visit. Note: Please advise the participant that for this questionnaire they are to interpret the instructions as referring to glasses or contacts they need for seeing objects at a distance (if required), not their reading glasses or bifocals.
* Photopic, high-contrast, best distance correction in the range of spherical -4.00 D to +1.00 D inclusively and cylinder < = + -2.00 D with photopic at the screening visit and photopic, high-contrast BCDVA of 20/25 or better OD and OS at the screening visit.
* Photopic, high-contrast HDVA of 20/32 or better OU at screening as well as before and 1 hour after dosing at both driving tests. Only monofocal correction (either spectacles or contact lenses) is allowed for the driving tests. If the participant does not have monofocal correction of 20/32 or better OU, the study site will provide monofocal spectacles.
* Mesopic, high-contrast DCNVA of 20/40 to 20/100 OD and OS at screening
* Photopic, high-contrast near visual acuity correctable to 20/40 or better in each eye at the screening visit.
* Mesopic pupil diameter < 8.0 mm in both eyes at the screening visit.

Exclusion Criteria:

* History of cataract surgery, phakic intraocular lens surgery, corneal inlay surgery, radial keratotomy, or any intraocular surgery.
* Use of any topical ophthalmic medications, including artificial tears other than the study medications during the study.
* Use of temporary or permanent punctal plugs or history of punctal cautery in one or both eyes.
* Corneal abnormalities in either eye that are likely to interfere with visual acuity.
* Narrow iridocomeal angles, history of angle-closure glaucoma, or previous iridotomy.
* Diagnosis of any type of glaucoma or ocular hypertension.
* Females who are pregnant, nursing, or planning a pregnancy during the study.
* Uncontrolled systemic disease.
* Severe dry eye disease.
* History of iris trauma.
* Lens opacity in either eye that is determined to cause significant disturbance of the central visual axis on screening biomicroscopy.

Ages: 40 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2021-05-14 (Actual); Primary Completion 2021-12-07 (Actual); Study Completion 2021-12-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (1):
- School of Optometry and Vision Science, Queensland University of Technology /ID# 226378, Brisbane, Queensland, Australia

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols, analyses plans, clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous independent scientific research, and will be provided following review and approval of a research proposal and statistical analysis plan and execution of a data sharing statement. Data requests can be submitted at any time after approval in the US and/or EU and a primary manuscript is accepted for publication. For more information on the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- [Derived] Waring GO 4th, Brujic M, McGee S, Micheletti JM, Zhao C, Schachter S, Liu H, Safyan E. Impact of presbyopia treatment pilocarpine hydrochloride 1.25% on night-driving performance. Clin Exp Optom. 2024 Aug;107(6):665-672. doi: 10.1080/08164622.2023.2279189. Epub 2023 Dec 3. PMID 38044272

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 43 participants were randomized and treated; 22 to the sequence AGN-190584 followed by vehicle and 21 to the sequence vehicle followed by AGN-190584.
Pre-assignment Details: The ITT population includes all randomized participants. The safety population includes all treated participants who received at least one dose of study intervention. All 43 randomized participants were included in both the intent-to-treat (ITT) and safety populations.
Groups:
- AGN-190584 - Vehicle (Sequence 1): Participants will receive AGN-190584 from Visit 2 through Visit 3 followed by Vehicle from Visit 4 through Visit 5.
- Vehicle - AGN-190584 (Sequence 2): Participants will receive Vehicle from Visit 2 through Visit 3 followed by AGN-190584 from Visit 4 through Visit 5.
Period: Period 1
Arm/Group | AGN-190584 - Vehicle (Sequence 1) | Vehicle - AGN-190584 (Sequence 2)
Started | 22 | 21
Completed | 22 | 21
Not Completed | 0 | 0
Period: Period 2
Arm/Group | AGN-190584 - Vehicle (Sequence 1) | Vehicle - AGN-190584 (Sequence 2)
Started | 22 | 21
Completed | 22 | 20
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: The ITT population includes all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | AGN-190584 - Vehicle (Sequence 1) | Vehicle - AGN-190584 (Sequence 2) | Total
Number analyzed (Participants) | 22 | 21 | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 22 | 21 | 43
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 50.9 (2.92) | 50.0 (4.22) | 50.5 (3.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 11 | 24
  Male | 9 | 10 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 22 | 21 | 43
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 1 | 2 | 3
  Black or African American | 1 | 0 | 1
  White | 18 | 19 | 37
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Composite Driving Z Score Approximately 1 Hour After Study Intervention Instillation
Description: An overall composite driving Z-score approximately 1 hour after study intervention instillation was derived to capture the overall driving performance of each participant compared with the whole group for the following parameters: percent hazards hit, percent sign recognition and recognition distance, pedestrian recognition distances, and percent of time outside of the lane. For each participant, the Z-score for each task of the driving test was the difference between his/her value and mean value of the assessments of all participants from the pooled data of both periods combined, divided by the standard deviation of all corresponding assessment values. Because a lower percentage of hazards hit, lower percentage of time outside of the driving lane, and a shorter lap duration indicate better driving performance, the Z-scores of these components were reversed (multiplied by -1) before computing the overall composite driving Z-score. A higher Z-score indicates better driving performance.
Time Frame: One hour after study intervention instillation at Visit 3 (Day 8 to 15) and at Visit 5 (Day 22 to 71)
Population: The ITT population includes all randomized participants. The primary efficacy endpoint was analyzed using a linear mixed-effects model with repeated measures (MMRM). Missing data were handled using an MMRM with the missing at random assumption, in which both missingness of data and the correlation of the repeated measurements were considered.
Measure: Mean (Standard Deviation); unit: Z-score
Groups:
- Vehicle; AGN-190584: In Sequence 1, participants received AGN-190584 from Visit 2 through Visit 3 followed by Vehicle from Visit 4 through Visit 5.
  In Sequence 2, participants received Vehicle from Visit 2 through Visit 3 followed by AGN-190584 from Visit 4 through Visit 5.
Arm/Group | Vehicle | AGN-190584
Number analyzed (Participants) | 43 | 42
Z-score | 0.118 (0.4011) | -0.121 (0.4503)
Statistical Analysis 1: Comparison: Vehicle vs AGN-190584; Test type: Non-Inferiority — Noninferiority of AGN-190584 was concluded if the lower bound of the 95% CI of the least-square mean difference between AGN-190584 and vehicle was greater than the pre-specified margin of -0.25; p = 0.0006, Mixed Models Analysis; Linear mixed-effects model with repeated measures; Least-Square (LS) Mean = -0.224, 95% CI 2-sided [-0.346 to -0.103], Standard Error of Mean 0.0602

2. Primary Outcome: Number of Participants With Adverse Events
Description: An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The investigator assesses the relationship of each event to the use of the study intervention. A serious adverse event (SAE) is an event that results in death, is life threatening, requires inpatient hospitalization or prolongs an existing hospitalization, results in a congenital anomaly, persistent or significant disability/incapacity or is an important medical event, that based on medical judgment, may jeopardize the participant and may require medical or surgical intervention to prevent any of the outcomes listed above.
Time Frame: Enrollment to Day 71
Population: The safety population includes all treated participants who receive ≥ 1 administration of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Vehicle | AGN-190584
Number analyzed (Participants) | 43 | 43
Participants | 8 | 32

ADVERSE EVENTS:
Time Frame: All-cause mortality and adverse event tables include events reported from enrollment to the end of the study. The median time participants were followed was 46 days for Period 1 (Vehicle); 37 days for Period 1 (AGN-190504); 8 days for Period 2 (Vehicle to AGN-190584); and 9 days for Period 2 (AGN-190584 to Vehicle).
Description: The safety population includes all participants who received at least one dose of study intervention. All 43 randomized participants were included in the safety population.
Groups:
- Period 1 (Vehicle): Participants received Vehicle from Visit 2 through Visit 3 in Period 1.
- Period 1 (AGN-190584): Participants received AGN-190584 from Visit 2 through Visit 3 in Period 1.
- Period 2 (Vehicle to AGN-190584): Participants received AGN-190584 from Visit 4 through Visit 5 in Period 2.
- Period 2 (AGN-190584 to Vehicle): Participants received Vehicle from from Visit 4 through Visit 5 in Period 2.
Arm/Group | Period 1 (Vehicle) | Period 1 (AGN-190584) | Period 2 (Vehicle to AGN-190584) | Period 2 (AGN-190584 to Vehicle)
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/22 | 0/21 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/22 | 0/21 | 0/22
Other Adverse Events (participants affected / at risk) | 2/21 | 14/22 | 15/21 | 3/22
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Period 1 (Vehicle) (N=21) | Period 1 (AGN-190584) (N=22) | Period 2 (Vehicle to AGN-190584) (N=21) | Period 2 (AGN-190584 to Vehicle) (N=22)
DRY EYE (Eye disorders) | 2 (4) | 1 (2) | 2 (3) | 1 (2)
EYE PAIN (Eye disorders) | 0 (0) | 2 (4) | 6 (12) | 0 (0)
OCULAR HYPERAEMIA (Eye disorders) | 0 (0) | 1 (2) | 2 (4) | 0 (0)
PHOTOPHOBIA (Eye disorders) | 0 (0) | 0 (0) | 2 (4) | 1 (2)
VISION BLURRED (Eye disorders) | 0 (0) | 4 (8) | 3 (6) | 1 (2)
VISUAL IMPAIRMENT (Eye disorders) | 0 (0) | 6 (14) | 6 (12) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
HEADACHE (Nervous system disorders) | 0 (0) | 5 (5) | 7 (7) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2021-10-28): https://cdn.clinicaltrials.gov/large-docs/82/NCT04837482/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-26): https://cdn.clinicaltrials.gov/large-docs/82/NCT04837482/SAP_001.pdf